CLINICAL TRIAL: NCT03786991
Title: EPI-STORM Cytokine Storm in Organ Donors: A Translational Study Linking Donor Epigenetic to Transplantation Success in Recipient
Brief Title: EPI-STORM: Cytokine Storm in Organ Donors
Acronym: EPI-STORM
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du CHUS (Unknown)
Responsible Party: Sponsor
Other Study IDs: MP-31-2019-2960
Record Dates: First submitted 2018-11-30; First posted 2018-12-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Organ Donation; Liver Transplantation; Kidney Transplantation; Graft Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (including miRNA and buffy coat) will be drawn at 5 specific time points: following ICU admission when patient has a serious neurological lesion, as soon as possible after consent to organ donation, as well as 4 to 8 hours and 24 hours after the first sample of phase 2 has been drawn. A final draw will be made prior to transfer from the ICU to operating room for organ recovery. A substudy will be conducted in some centers and we will collect samples at time of aortic cross clamp during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Organ donors: Organ donors after neurologic death (NDD) of 18 years old and older for whom consent to organ donation has been obtained.
  Interventions: Other: No intervention
- Liver and kidney Recipients: Liver and kidney recipients of 18 years old and older.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Kidney and liver transplantation are the treatment of choice and are often the last therapeutic option offered to patients with chronic renal and liver failure. More than 70% of kidneys and liver available for transplantation are obtained from donors following neurological death. Unfortunately, compared to living donation, transplant function, graft survival, and recipient survival are consistently inferior with kidneys and liver from neurologically deceased donors. This difference lies with the exacerbated pro-inflammatory state characteristic of deceased donors. Indeed, when neurologic death occurs, the immune system releases substances in the blood that could harm organs and particularly the liver and the kidneys. We believe that achieving a better understanding of the inflammatory processes of organ donors could be greatly informative to design future randomized controlled trial assessing the effect of personalized immunosuppressive therapy on organ donors to ultimately improve the care provided to donors so as to increase the number of organs available for transplantation and enhancing the survival of received grafts

DETAILED DESCRIPTION:
Severe neurological injuries, such as those observed in neurologically deceased donors, trigger a pro-inflammatory state that activates the immune system, increases vascular permeability, and recruits and activates immune cells in solid organs. The rapid and intense increase in circulating pro-inflammatory cytokines (e.g., IL-1, IL-6, TNF-α) following neurological death, has been referred to as the cytokine storm, one condition that is not seen among living donors. Interestingly, increased expression of TNF-α in the kidney and liver at the time of transplantation has been associated with reduced graft survival and acute rejection. Moreover, numerous studies have suggested that miRNA biomarkers can be targeted as diagnostic or therapeutic molecules in the field of organ transplantation. However, current models of graft injury fail to consider the epigenetic effects of physiological stressors that occurred in neurologically deceased donors. Although several biomarkers have been associated with graft dysfunction, the changes within the donor's inflammatory state, the mechanism underlying these events in donors, and the impacts on recipients are only poorly understood.

The investigators propose a multicenter prospective cohort study with the main objective of assessing the pro-inflammatory status of neurologically deceased donors by examining both miRNAs and circulatory cytokines and investigating its association with graft function in the recipient. Blood specimens will be collected at various time points in neurologically deceased liver and kidney donors in 5 organ recovery centres. The investigators hypothesize that in donors, Peak plasma concentration of pro-inflammatory cytokines and inflammatory-associated miRNAs targets (between consent and recovery) are associated with an increase in kidney delayed graft function and liver early graft dysfunction in the recipients. Considering that there is a therapeutic arsenal for treating donor cytokine storms( e.g., immunosuppressants) and that new targets based on a highly personalized mechanism could be developed we believe that the knowledge acquired in this research program will make it possible to improve the rate of livers and kidneys recovered from potential donors as well as enhance graft function in recipients.

ELIGIBILITY:
Phase 1 of the study:

Inclusion Criteria:

* Patient admitted to the intensive care unit with a serious neurologic lesion
* Glasgow Coma Scale score ≤ 4
* Absence of sedation for the last 6 hours
* Age ≥ 18 years old

Exclusion Criteria:

* S. aureus bacteremia
* Active neoplasia
* Receiving immunosuppressive therapy (including steroids) for > 3 months

Specific to potential liver donors:

* Hepatic insufficiency defined as i) INR > 1.5, ii) hepatic encephalopathy, iii) AST, ALT > 2 times normal value

Specific to potential kidney donors:

* Polycystic kidney disease
* Chronic renal failure (i.e., eGFR < 60 ml/min)

Phase 2 of the study:

Inclusion Criteria:

* Organ donor after neurologic death (DND) declaration as determined by the attending physician
* Consent to organ donation obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organ donors by neurologic death and liver and kidney recipients
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2018-12-16 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Kidney delayed graft function | 7-days post-transplantation
  Requirement for renal replacement therapy within the first 7 days following transplantation or decrease of < 10% of creatinine after 3 days after transplantation, or creatinine > 250 µmol/l at day 5 with evidence of delayed graft function by renal scintigraphy

SECONDARY OUTCOMES:
Liver early graft dysfunction | 7-days post-transplantation
  Presence of one of the following three criteria: (i) peak AST or ALT > 2000 U/L during the first 7 days, (ii) bilirubin ≥ 10 mg/dL on day 7 postoperatively, or (iii) INR ≥ 1.6 on day 7 postoperatively
Quantification of circulatory cytokines | From ICU admission up to organ recovery (5 timepoints(1:ICU admission; 2: consent to organ donation, 3: 4 to 8 hours after sample #2, 4: 24 hours after sample #2; 5: prior to transfer from ICU to operating room); 25 donors).
  Quantification of IL-1β, IL-2, IL-4, IL-6, IL-10, IL-12 (p70), IL-13, IFN-γ, and TNF-α by Luminex (Multiplex human cytokine panel, Millipore)
Identification of inflammatory-related miRNA targets using micro-transcriptome analyses | From ICU admission up to organ recovery (5 timepoints (1:ICU admission; 2: consent to organ donation, 3: 4 to 8 hours after sample #2, 4: 24 hours after sample #2; 5: prior to transfer from ICU to operating room) ;25 donors).
  Sequencing on an Illumina NovaSeq 6000 sequencing platform
Validation of inflammatory-related miRNA targets using targeted quantification | From ICU admission up to organ recovery (5 timepoints(1:ICU admission; 2: consent to organ donation, 3: 4 to 8 hours after sample #2, 4: 24 hours after sample #2; 5: prior to transfer from ICU to operating room); 105 donors).
  Quantification by RT-qPCR using TaqMan Advanced miRNA Assays
Validation of circulatory cytokines | From ICU admission up to organ recovery (5 timepoints (1:ICU admission; 2: consent to organ donation, 3: 4 to 8 hours after sample #2, 4: 24 hours after sample #2; 5: prior to transfer from ICU to operating room); 105 donors).
  Quantification of identified cytokines (in the 25 donors cohort) by Luminex (Multiplex, Millipore)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Frédérick D'Aragon, MD FRCPC MSc, Principal Investigator — Université de Sherbrooke
Locations (4):
- Canada (4):
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier Universitaire de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec- Université Laval, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clement AA, Lamarche D, Masse MH, Legare C, Tai LH, Fleury Deland L, Battista MC, Bouchard L, D'Aragon F. Time-course full profiling of circulating miRNAs in neurologically deceased organ donors: a proof of concept study to understand the onset of the cytokine storm. Epigenetics. 2022 Nov;17(11):1546-1561. doi: 10.1080/15592294.2022.2076048. Epub 2022 May 21. PMID 35603508